CLINICAL TRIAL: NCT06139029
Title: Comparison of 3% Normal Saline Nebulization Versus Steroid Nebulization in the Treatment of Bronchiolitis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mardan Medical Complex (Other)
Responsible Party: Principal Investigator, faizan sadiq, faizan sadiq,principal investigator, post graduate resident in pediatrics, Mardan Medical Complex
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 284/BKMC
Record Dates: First submitted 2023-11-04; First posted 2023-11-18 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Acute Bronchiolitis
Keywords: 3% normal saline; Bronchiolitis; Nebulization; Steroids.; Pediatric intensive care unit
MeSH Terms: conditions — Bronchiolitis | interventions — Saline Solution; Albuterol

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial was conducted at the Department of Pediatrics, Mardan Medical Complex, Mardan over a period of 4 months from 15th of November 2022 to 15th of March 2023.
  Sample size was calculated with OpenEpi calculator using 95% confidence level and power 80%.
  Estimated sample size 60, n1 (Patients in Group-A) =30, n2 (Patients in Group-B) =30.
  A total of 60 infants from both the genders between the ages of 3 to 12 months admitted in the pediatric unit with bronchiolitis were included in this study through non-probability consecutive sampling and equally randomized into 2 groups.
  Exclusion Criteria was set as infants having some underlying disease (e.g. Cystic fibrosis, bronchopulmonary dysplasia and cardiac or renal disease), prior history of wheezing, family history of asthma, pneumonia, TB, allergic history and progressive respira
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients in Group-A were nebulized with 3% normal saline (Experimental): Patients in Group-A were nebulized with 3% normal saline 3 times a day at intervals of 8 hours until they improved enough for discharge
  Interventions: Drug: 3% normal saline
- patients in Group-B were nebulized with steroid and salbutamol with 0.9% normal saline (Experimental): patients in Group-B were nebulized with steroid (beclomethasone dipropionate 400 μg/day in 3 divided doses) and salbutamol with 0.9% normal saline 3 times a day at intervals of 8 hours until they improved enough for discharge
  Interventions: Drug: steroid(beclomethasone dipropionate 400 μg/day) and salbutamol with 0.9% normal saline

INTERVENTIONS:
Drug: 3% normal saline — nebulization
  Arms: Patients in Group-A were nebulized with 3% normal saline
Drug: steroid(beclomethasone dipropionate 400 μg/day) and salbutamol with 0.9% normal saline — nebulization
  Arms: patients in Group-B were nebulized with steroid and salbutamol with 0.9% normal saline

SUMMARY:
To compare the efficacy of 3% normal saline nebulization and steroid nebulization in the treatment of bronchiolitis in infants.

DETAILED DESCRIPTION:
Comparison of 3% normal saline nebulization versus steroid nebulization in the treatment of bronchiolitis Abstract Objectives: To compare the efficacy of 3% normal saline nebulization and steroid nebulization in the treatment of bronchiolitis in infants.

Study Design: Randomized Controlled Trial Place and duration of study: This study was conducted at the Department of Pediatrics, Mardan Medical Complex, Mardan from 15th of November 2022 to 15th of March 2023.

Methods: A total of 60 infants between the ages of 3 to 12 months admitted in the pediatric unit with bronchiolitis were equally randomized into 2 groups. Patients in Group-A were nebulized with 3% normal saline while patients in Group-B were nebulized with steroid and salbutamol, 3 times a day at intervals of 8 hours until they improved enough for discharge. Assessment was done at 0, 12, 24, 48 and 72 hours using respiratory distress assessment instrument. Primary outcome was efficacy of the treatment defined as number of patients discharged from hospital in ≤ 72 hours after start of treatment. Efficacy between the 2 groups was compared by applying the chi-square test, p ≤0.05 was considered statistically significant.

Keywords: 3% normal saline, Bronchiolitis, Nebulization, Pediatric intensive care unit, Steroids.

Introduction:

Bronchiolitis is among the common acute infections reported at the pediatric units and is related to lower respiratory tract infections (RTI). These pediatric patients especially including infants are presented with signs of wheezing, crackles and mild to moderate breathing difficulties.The causes of bronchiolitis may include influenza (A & B), parainfluenza (A&B), adenovirus, human metapneumovirus, rhinovirus and coronavirus however the most common cause is reported to be respiratory syncytial virus (RSV). Bronchiolitis is a mild, self-limited infection in the majority of children but may sometimes progress to respiratory failure in infants.

The global prevalence of bronchiolitis is frequent and lower RTI caused by RSV was reported to be as high as 33 Million in 2019. A study collecting the data from intensive care registry of pediatrics in New Zealand and Australia reported an increase in admission rates due to bronchiolitis from 62.5 to 208 per 1,00,000 infants over a period of 12 years. In our region the RSV remains at its peak during the winter season and rainy seasons and is responsible for approximately 30 to 70% of the cases. This number is rising on yearly basis and the economic cost of the disease is also notable as the patients who required hospitalization was 3.6 Million and 26300 cases ended up to mortality. Every year, the cost of treating children with this condition is estimated to be in the millions of dollars.

The diagnosis of bronchiolitis is primarily based on the history and a rapid assay can detect the involvement of RSV. The symptoms of bronchiolitis typically begin with coughing and acute viral rhinitis. The infants then develop fever which may persist from 1 to 3 days and can lead to respiratory distress. The peak symptoms mostly appear in 4 four days which are related to maximum viral load, this duration however may vary among children. In severe cases, physical signs like inadequate nutrition and tachypnea are apparent which further appears in shape of chest hyperinflation, chest retractions, use of accessory muscles and decreased levels of SaO2. The presence of an elevated respiratory rate is a notable indicator of severity and apnea is an alert sign of developing respiratory failure.

Management of bronchiolitis includes the supportive interventions like oxygen and hydration which mostly helps to improve the course of disease while there is no specific treatment for infection is recommended. Infants reporting with symptoms of mild to moderate intensity are given the treatments including nasal saline, cool mist humidifier and paracetamol to control fever. The infants presenting with severity of symptoms like signs of dehydration and hypoxia and at risk of developing respiratory distress are recommended for immediate hospital admission. Interventions like aggressive hydration is important in these cases as their feeding is mostly compromised and the oxygen saturation must be kept above 90%. Treatments including beta-adrenergic agonists and steroids have been used in these cases however the efficacy data of these treatments is not decisive.

Methodology:

This randomized controlled trial was conducted at the Department of Pediatrics, Mardan Medical Complex, Mardan over a period of 4 months from 15th of November 2022 to 15th of March 2023.

Sample size was calculated with OpenEpi calculator using 95% confidence level and power 80%.

Expected efficacy in the treatment of bronchiolitis, P1 (3% normal saline nebulization) =94%, P2 (commonly used strategy) =58% .15 Estimated sample size 60, n1 (Patients in Group-A) =30, n2 (Patients in Group-B) =30.

A total of 60 infants from both the genders between the ages of 3 to 12 months admitted in the pediatric unit with bronchiolitis were included in this study through non-probability consecutive sampling and equally randomized into 2 groups.

Patients in Group-A were nebulized with 3% normal saline while patients in Group-B were nebulized with steroid (beclomethasone dipropionate 400 μg/day in 3 divided doses) and salbutamol with 0.9% normal saline, 3 times a day at intervals of 8 hours until they improved enough for discharge. Patients of both the groups will receive the supportive treatment as per needed including nasal suction, propped up position, organizing pneumonia (OP), intravenous (IV) fluid, oxygen therapy (when oxygen saturation <90%), paracetamol for fever, antibiotic, feeding and counseling.

Bronchiolitis was defined as when infant presenting with a rasping and persistent dry cough and noisy breathing (wheezing) with crackling or rattling sounds heard in the lungs on stethoscope on the respiratory distress assessment index (RDAI) with score of 4 to 15.

Patients were monitored by respiratory distress assessment instrument (RDAI) score initially at 0, 12, 24, 48 and 72 hours.

Efficacy was noted for both the groups on a given format. Primary outcome was efficacy of the treatment defined as number of patients discharged from hospital in ≤ 72 hours after start of treatment.

A written consent was taken from the parents/guardians of infants for the participation in study.

Permission for conducting study was taken from the ethical committee of the Hospital.

Data was analyzed using statistical analysis program SPSS 26. Mean ±SD was be calculated for quantitative variables like age, severity of bronchiolitis and duration of hospital stay. Frequencies and percentages were calculated for qualitative variables like gender and efficacy. Efficacy in between the 2 groups was compared by applying the chi-square test, where p ≤0.05 was considered statistically significant.

Discussion:

Bronchiolitis being the most common respiratory conditions in children and the most frequent reason of hospitalizations in infants under the age of 2 years has been frequently studied using different therapeutic options. During the past few years different researchers have mentioned the efficacy of 3% normal saline in comparison to other commonly used treatments in treating the bronchiolitis. Gupta V compared the efficacy of nebulization with 3% HS and 0.9% normal saline with salbutamol in infants with acute bronchiolitis. The clinical severity score of 3% HS solution as evaluated on 3rd day of treatment was 1.0 ± 1.1 compared clinical severity score of 3.3 ± 0.5 with 0.9% normal saline with salbutamol (p=0.000). The LHS was also significantly lower in 3% HS group compared to other group (3.4 ± 1.7 Vs 4.9 ± 1.4, p=0.001). The researchers thereby concluded that nebulization with 3% HS is not only effective but also help to cut the economic cost of treatment.

Stobbelaar K aimed to study the effects of nebulization with 3% HS in infants with an average age of 3.4 months admitted in the intensive care unit due to severe bronchiolitis. The results showed that nebulization with HS significantly reduced the need for respiratory support (P = 0.01) and LHS (P = 0.04) compared to patients who didn't received this treatment.

Majagaiya BS in their study conducted with infants suffering from moderate bronchiolitis compared the efficacy of nebulization with3% HS versus nebulization with 0.9% saline given 8 hourly, while salbutamol and corticosteroid was added to the therapies. The results of the study showed a significant improvement in CS score and decrease in LHS in the group taking 3% HS. The study thereby concluded that 3% HS solution is effective and safe choice for treating moderate bronchiolitis in infants.

In a recent study conducted in Pakistan, the comparison of efficacy was made between the group of infants taking the commonly recommended nebulization with salbutamol and other medications versus the group taking the HS nebulization for their bronchiolitis treatment. The CS score was significantly improved after 24 hours in the group taking 3% HS nebulization compared to group taking routine nebulization (p=0.000). Similarly LHS was significantly less in the group nebulized with HS (p=0.003).

Disclaimer of funding:

No

Conflict of interest:

No

Acknowledgments:

The services of departmental paramedic staff for their help in taking and keeping patient record are acknowledged.

ELIGIBILITY:
inclusion

1. age 3 to 12 months
2. both genders
3. acute brochiolitis as defined

exclusion

1. prior history of wheezing
2. family history of asthma
3. pneumonia
4. TB
5. progressive respiratory distress requiring mechanical ventillation
6. underlying diseases (e-g cystic fibrosis, bronchopulmonary dysplasia and cardiac or renal disease)

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
efficacy of 3% hypertonic saline in acute brochiolitis | discharged from hospital in ≤ 72 hours after start of treatment
  Primary outcome was efficacy of the treatment defined as number of patients discharged from hospital in ≤ 72 hours after start of treatment. Efficacy between the 2 groups was compared by applying the chi-square test, p ≤0.05 was considered statistically significant.

CONTACTS AND LOCATIONS:
Overall Officials: faizan sadiq, MBBS, Principal Investigator — Mardan Medical Complex
Locations (1):
- Faizan Sadiq, Mardan, Kpk, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: 2 weeks

REFERENCES:
- [Background] Stobbelaar K, Kool M, de Kruijf D, Van Hoorenbeeck K, Jorens P, De Dooy J, Verhulst S. Nebulised hypertonic saline in children with bronchiolitis admitted to the paediatric intensive care unit: A retrospective study. J Paediatr Child Health. 2019 Sep;55(9):1125-1132. doi: 10.1111/jpc.14371. Epub 2019 Jan 6. PMID 30645038
- [Background] Picone S, Fabiano A, Roma D, Di Palma F, Paolillo P. Re-comparing of three different epidemic seasons of bronchiolitis: different prophylaxis approaches. Ital J Pediatr. 2018 Dec 12;44(1):148. doi: 10.1186/s13052-018-0593-7. PMID 30541607
- [Background] Gold J, Hametz P, Sen AI, Maykowski P, Leone N, Lee DS, Gagliardo C, Hymes S, Biller R, Saiman L. Provider Knowledge, Attitudes, and Practices Regarding Bronchiolitis and Pneumonia Guidelines. Hosp Pediatr. 2019 Feb;9(2):87-91. doi: 10.1542/hpeds.2018-0211. Epub 2019 Jan 4. PMID 30610012
- [Background] Oz-Alcalay L, Ashkenazi S, Glatman-Freedman A, Weisman-Demri S, Lowenthal A, Livni G. Hospitalization for Respiratory Syncytial Virus Bronchiolitis in the Palivizumab Prophylaxis Era: Need for Reconsideration of Preventive Timing and Eligibility. Isr Med Assoc J. 2019 Feb;21(2):110-115. PMID 30772962
- [Background] Skjerven HO, Megremis S, Papadopoulos NG, Mowinckel P, Carlsen KH, Lodrup Carlsen KC; ORAACLE Study Group. Virus Type and Genomic Load in Acute Bronchiolitis: Severity and Treatment Response With Inhaled Adrenaline. J Infect Dis. 2016 Mar 15;213(6):915-21. doi: 10.1093/infdis/jiv513. Epub 2015 Oct 27. PMID 26508124
- [Background] Heppe Montero M, Gil-Prieto R, Walter S, Aleixandre Blanquer F, Gil De Miguel A. Burden of severe bronchiolitis in children up to 2 years of age in Spain from 2012 to 2017. Hum Vaccin Immunother. 2022 Dec 31;18(1):1883379. doi: 10.1080/21645515.2021.1883379. Epub 2021 Mar 2. PMID 33653212
- [Background] Panda S, Mohakud NK, Suar M, Kumar S. Etiology, seasonality, and clinical characteristics of respiratory viruses in children with respiratory tract infections in Eastern India (Bhubaneswar, Odisha). J Med Virol. 2017 Mar;89(3):553-558. doi: 10.1002/jmv.24661. Epub 2016 Aug 22. PMID 27509268
- [Background] Schlapbach LJ, Straney L, Gelbart B, Alexander J, Franklin D, Beca J, Whitty JA, Ganu S, Wilkins B, Slater A, Croston E, Erickson S, Schibler A; Australian & New Zealand Intensive Care Society (ANZICS) Centre for Outcomes & Resource Evaluation (CORE) and the Australian & New Zealand Intensive Care Society (ANZICS) Paediatric Study Group. Burden of disease and change in practice in critically ill infants with bronchiolitis. Eur Respir J. 2017 Jun 1;49(6):1601648. doi: 10.1183/13993003.01648-2016. Print 2017 Jun. PMID 28572120
- [Background] Li Y, Wang X, Blau DM, Caballero MT, Feikin DR, Gill CJ, Madhi SA, Omer SB, Simoes EAF, Campbell H, Pariente AB, Bardach D, Bassat Q, Casalegno JS, Chakhunashvili G, Crawford N, Danilenko D, Do LAH, Echavarria M, Gentile A, Gordon A, Heikkinen T, Huang QS, Jullien S, Krishnan A, Lopez EL, Markic J, Mira-Iglesias A, Moore HC, Moyes J, Mwananyanda L, Nokes DJ, Noordeen F, Obodai E, Palani N, Romero C, Salimi V, Satav A, Seo E, Shchomak Z, Singleton R, Stolyarov K, Stoszek SK, von Gottberg A, Wurzel D, Yoshida LM, Yung CF, Zar HJ; Respiratory Virus Global Epidemiology Network; Nair H; RESCEU investigators. Global, regional, and national disease burden estimates of acute lower respiratory infections due to respiratory syncytial virus in children younger than 5 years in 2019: a systematic analysis. Lancet. 2022 May 28;399(10340):2047-2064. doi: 10.1016/S0140-6736(22)00478-0. Epub 2022 May 19. PMID 35598608
- [Background] Fretzayas A, Moustaki M. Etiology and clinical features of viral bronchiolitis in infancy. World J Pediatr. 2017 Aug;13(4):293-299. doi: 10.1007/s12519-017-0031-8. Epub 2017 May 4. PMID 28470580
- [Background] Jo YM, Kim J, Chang J. Vaccine containing G protein fragment and recombinant baculovirus expressing M2 protein induces protective immunity to respiratory syncytial virus. Clin Exp Vaccine Res. 2019 Jan;8(1):43-53. doi: 10.7774/cevr.2019.8.1.43. Epub 2019 Jan 31. PMID 30775350
- [Background] Polack FP, Stein RT, Custovic A. The Syndrome We Agreed to Call Bronchiolitis. J Infect Dis. 2019 Jun 19;220(2):184-186. doi: 10.1093/infdis/jiz082. PMID 30783666